CLINICAL TRIAL: NCT02309658
Title: Safety and Efficacy of Gemcitabine Based Neoadjuvant Chemotherapy Followed by Chemoradiation in Locally Advanced Cervical Cancer Patients and Association With Human Equilibrative Nucleoside Transporter 1 (hENT1) Expression
Brief Title: Neoadjuvant Chemotherapy in Locally Advanced Cervical Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Carla Rameri Alexandre Silva de Azevedo, MD, Medical Oncologist, Professor Fernando Figueira Integral Medicine Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1156-1640
Record Dates: First submitted 2014-12-01; First posted 2014-12-05 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Cancer of Cervix
Keywords: cervix neoplasm; hENT1 protein, human; Chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Gemcitabine; Cisplatin; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional (Experimental): Treatment consisted of gemcitabine at a dose of 1000 mg/m2, followed by cisplatin 35 mg/m2 administered on day 1 and 8, for two cycles. After that, weekly cisplatin 40mg/m2 is administered concomitant with radiotherapy (45-55Gy) in 1,8-2,0 daily fractions and a 10Gy boost when there was parametrial involvement. Low-dose rate brachytherapy, in 4 fractions of 7Gy, in a total of 28Gy will complete the protocol.
  Interventions: Drug: gemcitabine; Drug: cisplatin; Radiation: chemoradiation

INTERVENTIONS:
Drug: gemcitabine — Patients received intravenous 500-1000 ml normal saline and antiemetic medication before chemotherapy. Treatment consisted of intravenous gemcitabine at a dose of 1000 mg/m2 diluted in 500 ml of normal saline administered over 30 minutes mg/m2 diluted in 500 ml of normal saline administered over 30 minutes on days 1 and 8, followed by cisplatin 35 mg/m2 administered over 2 hours on day 1 and 8.
  Other Names: Gemzar and cisplatin neoadjuvant chemotherapy
Drug: cisplatin — 35 mg/m2 administered over 2 hours on day 1 and 8.
Radiation: chemoradiation — external beam radiotherapy concomitant with weekly cisplatin 40mg/m2

SUMMARY:
The propose of this study is to determine if neoadjuvant chemotherapy followed by chemoradiation is safe and effective in locally advanced cervical cancer patients. Moreover, the study would determine if there is any association between hENT1 expression and response rate to gemcitabine.

DETAILED DESCRIPTION:
The study has been developed and executed at Medicina Integral Prof. Fernando Figueira Institute - IMIP since September/2013. The primary objective is to evaluate the safety of neoadjuvant chemotherapy based in gemcitabine followed by chemoradiation in cervical cancer patients. Data has been collected at medical oncology clinic, where patients have medical visits and receive chemotherapy treatment. New cases of cervical cancer patients are analysed for eligibility criteria. When matching these criteria, the protocol is explained, its participation is offered and consent form is explained, highlighting the voluntary aspect of the process. If there is agreement in participation, two consent forms are provided and signed. Patients receive one copy and the other one goes to his/her medical record. All demographic, social and medical data is recorded.

Patients are considered to have the first visit on the day they sign consent agreement form, when they are also referred to radiooncologist visit. Up to 30-business days they should complete staging (MRI, PET-SCAN, labs) and initiate neoadjuvant chemotherapy. Before each day, of each cycle, patients are seen by medical oncologist and nurse, when toxicity data is collected. Before and after neoadjuvant chemotherapy, there is a clinical evaluation performed by the gynecologic oncologist to evaluate clinical response. During chemoradiation, patients have weekly visits. The treatment is completed with brachytherapy, and 30-days after its completion, another clinical evaluation is done. After 90 days of completion treatment, pelvic MRI and PET-SCAN are repeated and considered to determine response rate.

Biopsies samples have been collected. The investigators intend to perform immunohistochemical analysis at the end of recruitment and identify any association between hENT1 expression and outcomes.

Information is collected by principal investigator in EXCEL forms, during medical visits. Toxicity data has been analyzed every 3 months by a data monitoring committee comprising two medical oncologists, one radiooncologist and a gynecological nurse. All unexpected event is related to this committee and also to the Research Ethics Committee of IMIP. Patients are followed up 3/3 months. Inconsistent or missing data will be re-checked in medical records.

This is a phase IIa study with only one arm of intervention. Since response rates observed in phase III studies with concomitant platin based chemoradiation is 85% in average, and given that response rate using gemcitabin based adjuvant chemotherapy, after chemoradiation, is 96.5%, the investigators calculated the sample size of 49 patients. It was considered an alpha error of 5% and 80% power. Descriptive analyses of variables of this population will be held. The normal numerical variables are described as mean +/- standard deviation. The non-parametric numeric variables are described as median (interquartile range). Categorical data will be described as a percentage of the total. The progression free survival and overall survival will be obtained by Kaplan-Meier method, using the computer program Epinfo.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed diagnostic of cervical carcinoma
* International Federation of Gynecology and Obstetrics (FIGO) stage Ib2 (>4cm) to IVa
* Performance status 0-2 (ECOG scale)
* Hemoglobin >10g/dl , neutrophil > 1500 /mm3, platelet >100.000/mm3
* Creatinine < 1,5 mg/dl
* Bilirubin total <1,6 mg/dl and liver enzymes (AST e ALT) < 2x (upper limit of normal)
* Informed consent.

Exclusion Criteria:

* Cervical tumors with adenocarcinoma, adenosquamous and small cell adenocarcinoma histology
* Distant metastasis including paraortic nodes
* Pregnancy and breast-feeding
* Previous chemotherapy, radiotherapy or uterine surgery
* Relevant co-morbidity which prevent chemotherapy use
* Previous neoplasia, except non-melanoma skin cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Toxicity will be evaluated with Common Terminology Criteria for Adverse Events (CTCAE 4,0). | Up to 4 weeks after brachytherapy
  Toxicity will be recorded before each day of chemotherapy and weekly during radiotherapy.
Response rate (Response Evaluation Criteria in Solid Tumors (RECIST) criteria with pelvic MRI and PET-CT) | 12 weeks after treatment
  Response will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) criteria with pelvic MRI and PET-CT.
  Immediately after neoadjuvant chemotherapy and 30 days after brachytherapy, clinical response will also be evaluated.

SECONDARY OUTCOMES:
Disease free survival | One year of follow up.
  From recruitment date to relapse date.
Overall Survival | One year of follow up.
  From recruitment date to death.
hENT1 expression | At the end of recruitment, expected to be at 24 months after study beginning
  hENT1 will be analysed by immunohistochemistry. Scoring for hENT1 was based on staining intensities and the proportion of cancer cells. Islet cells of pancreas tissue served as an external positive control for hENT1 immunohistochemistry, and lymphocytes or endothelial cells surrounding the tumour area served as internal positive controls. Carcinoma was then evaluated by comparison with the internal controls. Staining intensity was graded as: 0, absent; 1+, positive but less intense than internal control tissue; 2+, positive as in internal control tissue; and 3+,positive, more intense than internal control tissue. Samples with regions of varying staining intensities of hENT1 were scored and the percentages of each region were recorded. Finally, tumours with an intensity staining of 3+in≥50% of the tumour cells were considered as showing high expression of hENT1.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Rameri A. de Azevedo, MD, Principal Investigator — IMIP
Locations (1):
- Instituto de Medicina Integral Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Chemoradiotherapy for Cervical Cancer Meta-Analysis Collaboration. Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data from 18 randomized trials. J Clin Oncol. 2008 Dec 10;26(35):5802-12. doi: 10.1200/JCO.2008.16.4368. Epub 2008 Nov 10. PMID 19001332
- [Background] Eifel PJ, Winter K, Morris M, Levenback C, Grigsby PW, Cooper J, Rotman M, Gershenson D, Mutch DG. Pelvic irradiation with concurrent chemotherapy versus pelvic and para-aortic irradiation for high-risk cervical cancer: an update of radiation therapy oncology group trial (RTOG) 90-01. J Clin Oncol. 2004 Mar 1;22(5):872-80. doi: 10.1200/JCO.2004.07.197. PMID 14990643
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Kies MS, Haraf DJ, Athanasiadis I, Kozloff M, Mittal B, Pelzer H, Rademaker AW, Wenig B, Weichselbaum RR, Vokes EE. Induction chemotherapy followed by concurrent chemoradiation for advanced head and neck cancer: improved disease control and survival. J Clin Oncol. 1998 Aug;16(8):2715-21. doi: 10.1200/JCO.1998.16.8.2715. PMID 9704722
- [Background] Whitney CW, Sause W, Bundy BN, Malfetano JH, Hannigan EV, Fowler WC Jr, Clarke-Pearson DL, Liao SY. Randomized comparison of fluorouracil plus cisplatin versus hydroxyurea as an adjunct to radiation therapy in stage IIB-IVA carcinoma of the cervix with negative para-aortic lymph nodes: a Gynecologic Oncology Group and Southwest Oncology Group study. J Clin Oncol. 1999 May;17(5):1339-48. doi: 10.1200/JCO.1999.17.5.1339. PMID 10334517
- [Background] Rose PG, Bundy BN, Watkins EB, Thigpen JT, Deppe G, Maiman MA, Clarke-Pearson DL, Insalaco S. Concurrent cisplatin-based radiotherapy and chemotherapy for locally advanced cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1144-53. doi: 10.1056/NEJM199904153401502. PMID 10202165
- [Background] Pearcey R, Brundage M, Drouin P, Jeffrey J, Johnston D, Lukka H, MacLean G, Souhami L, Stuart G, Tu D. Phase III trial comparing radical radiotherapy with and without cisplatin chemotherapy in patients with advanced squamous cell cancer of the cervix. J Clin Oncol. 2002 Feb 15;20(4):966-72. doi: 10.1200/JCO.2002.20.4.966. PMID 11844818
- [Background] Neoadjuvant Chemotherapy for Locally Advanced Cervical Cancer Meta-analysis Collaboration. Neoadjuvant chemotherapy for locally advanced cervical cancer: a systematic review and meta-analysis of individual patient data from 21 randomised trials. Eur J Cancer. 2003 Nov;39(17):2470-86. doi: 10.1016/s0959-8049(03)00425-8. PMID 14602133
- [Background] Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1137-43. doi: 10.1056/NEJM199904153401501. PMID 10202164
- [Result] Duenas-Gonzalez A, Rivera L, Mota A, Lopez-Graniel C, Guadarrama A, Gonzalez A, Chanona G, Cabrera P, de la Garza J. The advantages of concurrent chemoradiation after neoadjuvant chemotherapy for locally advanced cervical carcinoma. Arch Med Res. 2002 Mar-Apr;33(2):201-2. doi: 10.1016/s0188-4409(01)00358-7. No abstract available. PMID 11886723
- [Result] Duenas-Gonzalez A, Lopez-Graniel C, Gonzalez A, Reyes M, Mota A, Munoz D, Solorza G, Hinojosa LM, Guadarrama R, Florentino R, Mohar A, Melendez J, Maldonado V, Chanona J, Robles E, De la Garza J. A phase II study of gemcitabine and cisplatin combination as induction chemotherapy for untreated locally advanced cervical carcinoma. Ann Oncol. 2001 Apr;12(4):541-7. doi: 10.1023/a:1011117617514. PMID 11398890
- [Result] Matsumura N, Nakamura Y, Kohjimoto Y, Inagaki T, Nanpo Y, Yasuoka H, Ohashi Y, Hara I. The prognostic significance of human equilibrative nucleoside transporter 1 expression in patients with metastatic bladder cancer treated with gemcitabine-cisplatin-based combination chemotherapy. BJU Int. 2011 Jul;108(2 Pt 2):E110-6. doi: 10.1111/j.1464-410X.2010.09932.x. Epub 2010 Dec 16. PMID 21166756
- [Result] Giovannetti E, Del Tacca M, Mey V, Funel N, Nannizzi S, Ricci S, Orlandini C, Boggi U, Campani D, Del Chiaro M, Iannopollo M, Bevilacqua G, Mosca F, Danesi R. Transcription analysis of human equilibrative nucleoside transporter-1 predicts survival in pancreas cancer patients treated with gemcitabine. Cancer Res. 2006 Apr 1;66(7):3928-35. doi: 10.1158/0008-5472.CAN-05-4203. PMID 16585222
- [Result] Duenas-Gonzalez A, Zarba JJ, Patel F, Alcedo JC, Beslija S, Casanova L, Pattaranutaporn P, Hameed S, Blair JM, Barraclough H, Orlando M. Phase III, open-label, randomized study comparing concurrent gemcitabine plus cisplatin and radiation followed by adjuvant gemcitabine and cisplatin versus concurrent cisplatin and radiation in patients with stage IIB to IVA carcinoma of the cervix. J Clin Oncol. 2011 May 1;29(13):1678-85. doi: 10.1200/JCO.2009.25.9663. Epub 2011 Mar 28. PMID 21444871
- [Result] Borbath I, Verbrugghe L, Lai R, Gigot JF, Humblet Y, Piessevaux H, Sempoux C. Human equilibrative nucleoside transporter 1 (hENT1) expression is a potential predictive tool for response to gemcitabine in patients with advanced cholangiocarcinoma. Eur J Cancer. 2012 May;48(7):990-6. doi: 10.1016/j.ejca.2011.11.006. Epub 2011 Dec 1. PMID 22137164